CLINICAL TRIAL: NCT02021942
Title: Efficacy of Medical Treatment With SOM230 LAR in Patients With Primary Inoperable Thymoma and/or With Local Recurrent Thymoma to Reduce Tumor Size
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Prof. Dr. Berthold Schalke (Other)
Collaborators: Crolll Gmbh (Other)
Responsible Party: Sponsor-Investigator, Prof. Dr. Berthold Schalke, Prof. Dr. Berthold Schalke, University of Regensburg
Organization: University of Regensburg (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CSOM230CIC01T
Record Dates: First submitted 2013-12-20; First posted 2013-12-27 (Estimated); Results first posted 2018-02-05 (Actual); Last update posted 2018-02-05 (Actual); Status verified 2017-07

CONDITIONS: Primary Inoperable Thymoma; Local Recurrent Thymoma
Keywords: primary inoperable thymoma; local recurrent thymoma; reduction of tumor size; SOM230 LAR
MeSH Terms: interventions — pasireotide; Octreotide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- SOM230 LAR (Experimental): SOM230 LAR in a dosage of 60 mg i.m. once every 4 weeks
  Interventions: Drug: SOM230 LAR

INTERVENTIONS:
Drug: SOM230 LAR — SOM230 LAR in a dosage of 60 mg is administered i.m. once every 4 weeks.
  Other Names: Pasireotide; Sandostatin®

SUMMARY:
This is a monocenter, single-arm, open label phase II trial evaluating the effect of SOM230 LAR in adult patients with inoperable primary thymoma and thymoma metastasis (Masaoka II-IVa). SOM230 LAR in a dosage of 60 mg is administered i.m. once every 4 weeks. The purpose of this trial is a proof of concept.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients aged ≥18 years
* Diagnosis of thymoma as assessed by biopsy and/or szintigraphy
* Inoperability of thymoma or loco-regional metastases. Inoperability is defined as at least adherence of the tumor to the neighbored organs, suspicious to infiltrate neighbored organs or local metastasis so that R0 resection can not be expected and /or local recurrence of thymic tumor
* Tumor stage: Thymomas of all WHO based histological subtypes (WHO A, AB, B1, B2, B3) (Rosai, 1999; Travis 2004) at Masaoka stage II to IVa based on histological examination of resection specimens or core biopsies.
* Patients with and without thymoma associated paraneoplastic syndrome.
* Performance status 0,1, or 2 (ECOG)
* Patients for whom written informed consent to participate in the study has been obtained

Exclusion Criteria:

* Patients having received radiolabeled somatostatin analogue therapy within the 6 months or any cytotoxic chemotherapy or interferon therapy within the 2 months prior to recording baseline symptoms
* Patients who have undergone major surgery/surgical therapy for any cause within 1 month or surgical therapy of loco-regional metastases within the last 3 months before recording baseline symptoms
* Patients who have received radiotherapy for any reason within the last 4 weeks and must have recovered from any side effects of radiotherapy before recording baseline symptoms
* Patients who are not biochemically euthyroid
* Diabetic patients on antidiabetic medications whose fasting blood glucose is poorly controlled as indicated by HbA1C > 8%
* Patients with symptomatic cholelithiasis
* Patients who have congestive heart failure (NYHA Class III or IV), unstable angina, sustained ventricular tachycardia, ventricular fibrillation, clinically significant bradycardia, advanced heart block or a history of acute myocardial infarction within the six months preceding enrollment
* Patients with QT related risk factor: QTcF at screening > 450 msec
* Patients with QT related risk factor: History of syncope or family history of idiopathic sudden death
* Patients with QT related risk factor:Sudden or clinically significant cardiac arrhythmias
* Patients with QT related risk factor: Risk factors for Torsades de Pointes such as hypokalemia, hypomagnesemia, cardiac failure, clinically significant / symptomatic bradycardia, or high-grade AV block
* Patients with QT related risk factor: Concomitant disease(s) that could prolong QT such as autonomic neuropathy (caused by diabetes or Parkinson's disease), HIV, cirrhosis, uncontrolled hypothyroidism or cardiac failure
* Patients with QT related risk factor: Concomitant medication(s) known to increase the QT interval
* Patients with potassium <3.0 mmol/L at study entry, magnesium <0.4 mmol/L at study entry, calcium <1.75 mmol/L at study entry, family history of long QT syndrome, and concomitant medications known to prolong the QT interval. If the electrolyte abnormalities are corrected prior to study commencement, the patient may become eligible for the trial.
* Patients with liver disease such as cirrhosis, chronic active hepatitis or chronic persistent hepatitis with serum bilirubin > 1.5 X ULN, serum albumin < 0.67 X LLN, and/or ALT or AST more than 2 X ULN for patients without liver Confidential - 20 - Amended Clinical Study Protocol v01 / Track Changes Study No. CSOM230CIC01T metastases or ALT or AST more than 5X ULN for patients with documented liver metastases
* Patients with additional active malignant disease within the last five years (with the exception of basal cell carcinoma or carcinoma in situ of the cervix)
* Patients with the presence of active or suspected acute or chronic uncontrolled infection or with a history of immunocompromise, including a positive HIV test result (ELISA and Western blot). A HIV test will not be required; however, previous medical history will be reviewed
* Patients with abnormal coagulation (PT or APTT elevated by 30% above normal limits)
* Patients with WBC <2.5 X 109/L; Hgb <10 g/dL; PLT <100 X 109/L (patients with paraneoplastic pan-, leuco-, erythro- or thrombopenia can be included if this seems to be the only reason for pan-, leuco-, erythro- or thrombopenia)
* Known hypersensitivity to somatostatin analogues or any component of the pasireotide or octreotide LAR or s.c. formulations
* Patients who have any current or prior medical condition that may interfere with the conduct of the study or the evaluation of its results in the opinion of the investigator
* Female patients who are pregnant or lactating, or are of childbearing potential and not practicing a medically acceptable method of birth control. Female patients must use a secure method of contraception if sexually active and the partner should use a condom. If oral contraception is used, the patient must have been practicing this method for at least two months prior to enrollment and must agree to continue the oral contraceptive throughout the course of the study, and for three months after the study has ended. Male patients who are sexually active are required to use condoms during the study and for three months afterwards as a precautionary measure (available data do not suggest any increased reproductive risk with the study drugs). Female partners of these male patients should use a secondary barrier contraception.
* Patients who are currently part of or have participated in any clinical investigation with an investigational drug within 1 month prior to dosing
* Patients with a history of non-compliance to medical regimens or who are considered potentially unreliable or will not be able to complete the entire study
* Patient has received any other investigational agents within 28 days of first day of study drug dosing
* Abnormal clinical laboratory values considered by the investigator to be clinically significant and which could affect the interpretation of the study results

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2012-03; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Berthold Schalke, Prof. Dr., Principal Investigator — Professor
Locations (1):
- Klinik und Poliklinik für Neurologie der Universität Regensburg, Regensburg, Bavaria, Germany

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This monocentric trial was conducted in Regensburg, Germany. The patients were asked for study participation by the investigator.
Period: Overall Study
Arm/Group | SOM230 LAR
Started | 16
Completed | 16
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | SOM230 LAR
Number analyzed (Participants) | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.6 (12.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 9
Region of Enrollment [Count of Participants; unit: Participants]
  Germany | 16

OUTCOME MEASURES:

1. Primary Outcome: Percent Change in Tumor Volume From Baseline to EOS
Description: To evaluate whether SOM230 LAR is effective in patients with inoperable thymoma with respect to shrinkage of tumor volume. Response is defined as the decrease in tumor volume of 20 % at EOS as compared to baseline. Tumor shrinkage is assessed by CT or MRI.
Time Frame: at least 6 months
Population: Initial diagnosis of thymoma for one patient could not be confirmed, but a squamous cell carcinoma was diagnosed by the central pathologist. Tumor voume was 320.99 cm^3 at screening. Tumor size was reduced to 176.87 cm^3 at month 2 (-44.9 % compared to baseline). At month 4 (EOS) tumor volume was slightly increased compared to month 2 (189 cm^3).
Measure: Mean (95% Confidence Interval); unit: percentage of tumor volume
Arm/Group | SOM230 LAR
Number analyzed (Participants) | 16
percentage of tumor volume | -37.38 [-60.88 to -13.88]

2. Secondary Outcome: Tumor Resection Status
Description: To evaluate the resection status based on the categories R0, R1 and ≥ R2 at EOS using CT or MRI imaging.
  R0 resection means no residual tumor tissue (best status); R1 indicates microscopic residual tumor tissue and R2 indicates macroscopic residual tumor tissue (worst status).
Time Frame: at least 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | SOM230 LAR
Number analyzed (Participants) | 16
Participants
  Surgery performed with resection status R0 | 6
  Surgery performed with resection status R1 | 4
  No surgery performed | 6

3. Secondary Outcome: Assessment of Tumor Operability
Description: Assessment if patients reaching operability at the EOS.
Time Frame: at least 6 months
Population: Operability of the tumor at the EOS was based on the decision of the treating surgeon. In addition the response criteria had to be fulfilled.
  The tumors of 11 patients (68.75%) were operable. One of these patients decided not to undergo surgery. Tumors of 5 patients were inoperable (31.25%) at the EOS.
Measure: Count of Participants; unit: Participants
Arm/Group | SOM230 LAR
Number analyzed (Participants) | 16
Participants
  Tumor assesed as operable. | 11
  Tumor assesed as not operable. | 5

4. Other Pre Specified Outcome: Safety: Number of Participants With Adverse Events (AE) and Serious Adverse Events (SAE)
Time Frame: at least 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | SOM230 LAR
Number analyzed (Participants) | 16
Participants
  Number of participants with AEs | 16
  Number of participants with SAEs | 7

5. Other Pre Specified Outcome: Assessment of Myasthenia Gravis (MG) Status by Determining Titin-antibody Status
Description: MG severity status is assessed by determining Titin-antibody status at Baseline and EOS.
Time Frame: at least 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | SOM230 LAR
Number analyzed (Participants) | 16
Participants
  Missing data at baseline or EOS | 8
  Change from negative to negative | 4
  Change from negative to positive | 0
  Change from positive to positive | 2
  Change from positive to negative | 2

6. Other Pre Specified Outcome: Assessment of Myasthenia Gravis (MG) Status by Measuring ACHR-antibody Concentrations
Description: MG severity status is assessed by measuring ACHR-antibody concentrations at Baseline and EOS.
Time Frame: at least 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | SOM230 LAR
Number analyzed (Participants) | 16
Participants
  Missing data at baseline or EOS | 8
  ACHR-antibody level increased | 1
  ACHR-antibody level decreased | 4
  ACHR-antibody level constant | 3

7. Other Pre Specified Outcome: Health Related Quality of Life
Description: Health related quality of life information was collected at Baseline and EOS using SF-36 questionnaire. Questionnaires had to be completed by the patients. All questions are scored on a scale from 0 to 100, with 100 representing the highest level of functioning possible.
  Patient reported answers were transformed into domain scores according to the guidelines provided by RAND/MOS. Statistical significance of the result was tested with a paired Wilcoxon rang sum test with a significance level of 0.05 considering only paired values (n=11) using PSPP Version 0.10.1.
Time Frame: at least 6 months
Population: 5 out of 16 patients were excluded from analysis due to missing EOS data.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | SOM230 LAR
Number analyzed (Participants) | 11
units on a scale
  Physical function (SCR) | 58.6 (28.9)
  Physical function (EOS) | 49.1 (25.6)
  Role limitations due to physical health (SCR) | 31.8 (38.9)
  Role limitations due to physical health (EOS) | 34.1 (45.1)
  Pain (SCR) | 57.3 (28.8)
  Pain (EOS) | 52.3 (35.7)
  General health (SCR) | 53.2 (12.9)
  General health (EOS) | 47.1 (14.5)
  Energy/Fatigue (SCR) | 43.6 (15.5)
  Energy/Fatigue (EOS) | 39.2 (21.3)
  Social functioning (SCR) | 61.4 (27.6)
  Social functioning (EOS) | 60.2 (30.5)
  Role limitations due to emotional problems (SCR) | 63.6 (45.8)
  Role limitations due to emotional problems (EOS) | 60.6 (44.3)
  Emotional well-being (SCR) | 60.4 (18.7)
  Emotional well-being (EOS) | 56.6 (20.9)
  Change in health (general) (SCR) | 38.6 (20.5)
  Change in health (general) (EOS) | 50.0 (15.8)

ADVERSE EVENTS:
Time Frame: Baseline, i.e. start of study drug, through study completion (EOS, including four weeks following the last dose of study drug).
Description: An adverse event (AE) is the appearance or worsening of any undesirable sign, symptom, or medical condition occurring after starting the study drug even if the event is not considered to be related to study drug. Medical conditions/diseases present before starting study drug are only considered AE if they worsen after starting study drug.
Arm/Group | SOM230 LAR
All-Cause Mortality (participants affected / at risk) | 0/16
Serious Adverse Events (participants affected / at risk) | 7/16
Other Adverse Events (participants affected / at risk) | 16/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SOM230 LAR (N=16)
Anaemia (Blood and lymphatic system disorders) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (1)
Systemic inflammatory response syndrome (General disorders) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Foot fracture (Injury, poisoning and procedural complications) | 1 (1)
Spinal fracutre (Injury, poisoning and procedural complications) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 3 (3)
Metastasis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Embolism (Vascular disorders) | 1 (1)
Venous thrombosis (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SOM230 LAR (N=16)
Leukocytosis (Blood and lymphatic system disorders) | 3 (3)
Cushing's syndrome (Endocrine disorders) | 1 (1)
Cataract (Eye disorders) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 10 (12)
Abdominal pain (Gastrointestinal disorders) | 3 (4)
Vomiting (Gastrointestinal disorders) | 2 (2)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1)
Abnormal faeces (Gastrointestinal disorders) | 1 (1)
Flatulence (Gastrointestinal disorders) | 1 (1)
Haemorrhoids (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Oral dysaesthesia (Gastrointestinal disorders) | 1 (1)
Chest pain (General disorders) | 3 (3)
Fatigue (General disorders) | 1 (1)
Influenza like illness (General disorders) | 1 (1)
Malaise (General disorders) | 1 (1)
Oedema peripheral (General disorders) | 1 (1)
Peripheral swelling (General disorders) | 1 (1)
Pyrexia (General disorders) | 1 (1)
Immunodeficiency (Immune system disorders) | 1 (1)
Cystitis (Infections and infestations) | 2 (2)
Nasopharyngitis (Infections and infestations) | 2 (2)
Skin infection (Infections and infestations) | 2 (2)
Bacterial infection (Infections and infestations) | 1 (1)
Oral candidiasis (Infections and infestations) | 1 (1)
Oral herpes (Infections and infestations) | 1 (1)
Penile infection (Infections and infestations) | 1 (1)
Vaginal infection (Infections and infestations) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 1 (1)
Muscle strain (Injury, poisoning and procedural complications) | 1 (1)
Gamma-glutamyltransferase increased (Investigations) | 2 (2)
Blood creatine phosphokinase increased (Investigations) | 1 (1)
Glycosylated haemoglobin increased (Investigations) | 1 (1)
Troponin increased (Investigations) | 1 (1)
Weight decreased (Investigations) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 4 (12)
Diabetes mellitus (Metabolism and nutrition disorders) | 2 (2)
Gout (Metabolism and nutrition disorders) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 3 (3)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
Dysgeusia (Nervous system disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1)
Glycosuria (Renal and urinary disorders) | 1 (1)
Haematuria (Renal and urinary disorders) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Laryngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 (1)
Flushing (Vascular disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Eval. of 3 intended secondary efficacy parameters was suspended due to scarcity of resources:

histopath. eval. of tumor samples, immunohistochem. eval. of tumor derived cells and eval. of changes in the subset composition of intratumorous T-cells

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes